CLINICAL TRIAL: NCT00205049
Title: A Pilot Study of Pentoxifylline-Therapy for Acute Alcoholic Hepatitis
Brief Title: Pentoxifylline for Acute Alcoholic Hepatitis (AAH)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of funding
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: M-2004-0388
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-04

CONDITIONS: Hepatitis, Alcoholic
Keywords: acute alcoholic hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pentoxifylline/Placebo (Experimental): All subjects will be randomized to receive either pentoxifylline 400mg orally or placebo 3 times daily for 28 days (20-40 treated, 1-20 placebo) with monthly follow up for 90 days.
  Interventions: Drug: pentoxifylline

INTERVENTIONS:
Drug: pentoxifylline — daily dosing
  Other Names: no other names

SUMMARY:
The goal of this study is to demonstrate the effectiveness of pentoxifylline compared to placebo in AAH while studying putative mechanisms that are plausible and testable. The main hypothesis is that pentoxifylline reduces the 90-day mortality of AAH.

DETAILED DESCRIPTION:
The goal of this study is to demonstrate the effectiveness of pentoxifylline compared to placebo in AAH while studying putative mechanisms that are plausible and testable. The main hypothesis is that pentoxifylline reduces the 90-day mortality of AAH.

This study never moved forward due to funding issues.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient with acute alcoholic hepatitis
* Model for End-Stage Liver Disease (MELD) of 15 or greater
* Recent alcohol abuse

Exclusion Criteria:

* Recent infection
* Other life threatening disease
* Severe coagulopathy
* Another non-alcoholic cause of liver disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2005-03; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Lucey, MD, Principal Investigator — University of Wisconsin, Madison

RESULTS

PARTICIPANT FLOW:
Groups:
- Pentoxifylline; Placebo: All subjects will be randomized to receive either pentoxifylline 400mg orally or placebo 3 times daily for 28 days
Period: Overall Study
Arm/Group | Pentoxifylline | Placebo
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pentoxifylline | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants]
Sex/Gender, Customized [Number; unit: 0]

OUTCOME MEASURES:

1. Primary Outcome: Survival at 28 Days
Time Frame: 28 days
Population: Study was terminated before any data was gathered/analyzed.
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Pentoxifylline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study was terminated before any data was gathered/analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No